CLINICAL TRIAL: NCT05432661
Title: clınıcal Effects of High-flow Nasal Oxygen Use ın gerıatrıc patıents usıng Endoscopic Retrograde Cholangiopancreatography Under sedatıon
Brief Title: clınıcal Effects of High-flow Nasal Oxygen Use ın gerıatrıc patıents
Acronym: HFNO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yunus Emre (Other)
Responsible Party: Sponsor-Investigator, Yunus Emre, SPECIALIST DOCTOR, Ankara Training and Research Hospital
Organization: Ankara Training and Research Hospital (Other)
Other Study IDs: ytuncdemir
Record Dates: First submitted 2022-06-13; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Biliary Obstruction; Oddi's Sphincter Constriction; Biliary Stones
Keywords: nasal oxygen; high flow nasal oxygen; geriatric; endoskopic retrograde cholangiopancreatography
MeSH Terms: conditions — Cholecystolithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1 nasal kanul: The data of a total of 60 patients in the group will be recorded. Those with saturation below 92% will be included in the study. The data of the nasal cannula group will be obtained from retrospective file and archive scanning. After providing standard monitoring, preoxygenation was performed for 3 minutes. After preoxygenation, 2-4 L/min oxygen was given to the patients who would receive oxygen support by nasal cannula. Patients were followed for at least 15 minutes after the procedure or until the patient recovered. Our aim is the early recovery of patients without complications.
- 2 HİGH-FLOW NASAL OXYGEN: The data of a total of 60 patients in the group will be recorded. Those with saturation below 92% will be included in the study. After the standard monitoring is established, preoxygenation will be performed for 3 minutes. . After preoxygenation, 40 L/min oxygen will be administered through a HFNO system to patients who will receive oxygen support with HFNO ( Inspired O2 FLO High Flow Oxygen Therapy ). Patients will be followed for a minimum of 15 minutes after the procedure or until the patient recovers.
  Interventions: Device: HİGH-FLOW NASAL OXYGEN USE (HFNO)

INTERVENTIONS:
Device: HİGH-FLOW NASAL OXYGEN USE (HFNO) — It is aimed to show that the use of HFNO can improve oxygenation compared to the use of nasal cannula in ERCP procedures performed under sedation in the prone position.
  Groups: 2 HİGH-FLOW NASAL OXYGEN

SUMMARY:
It is designed to monitor the efficacy of nasal cannula or hıgh-flow nasal oxygen in geriatric patients for endoscopıc retrograde cholangıopancreatography procedures. The aim of the study is to evaluate the efficacy and safety of oxygen support obtained with low-flow nasal cannula and hıgh-flow nasal oxygen during endoscopıc retrograde cholangıopancreatography in the patient group at risk for adverse respiratory events. We hypothesized that high-flow nasal oxygen administration can prevent adverse respiratory events such as deep sedation and patient position that may endanger the airway safety of patients, and reduce the problems in cardiac and hemodynamic parameters that may develop.

DETAILED DESCRIPTION:
In this retroprospective study, it was aimed to compare the effects of high flow nasal oxygen and standard nasal cannula use on hypoxia and oxygenation in geriatric endoscopic retrograde cholangiopancreatography cases performed under sedation in the prone position. Data belonging to the nasal cannula group will be obtained by scanning the forms and files retrospectively. Data in the high flow nasal oxygen group will be prospectively recorded during the procedure.

After the general anesthesia approval of the patients who will be applied ERCP, they are taken to the application room in the endoscopy unit. Here, standard monitoring (pulse oximetry, electrocardiography (ECG), non-invasive blood pressure measurement) is performed according to the criteria of the American Society of Anesthesiologists (ASA). in sedated patients for endoscopic retrograde cholangiopancreatography intervention, starting 5 minutes before sedation at 5-minute intervals; During the application, blood pressure, pulse, SpO2, presence of arrhythmia, interruptions due to airway interventions are monitored by the anesthesiologist and recorded in the case report form.

After the standard monitoring is established, preoxygenation is performed for 3 minutes. Then, 5 L/min of oxygen is given through the nasal cannula throughout the procedure. Patients who will receive oxygen support with high flow nasal oxygen (Inspired O2 FLO High Flow Oxygen Therapy) will be given 40 L/min oxygen with a high flow nasal oxygen system after preoxygenation. Patients will be followed for at least 15 minutes after the procedure or until the patient recovers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with physical condition class II-III of the American Society of Anesthesiologists, ----aged 65-90,
* with Spo2 of 92% and/or below in room air,

Exclusion Criteria:

Coagulation disorder, nasopharyngeal obstruction,

* bleeding tendency,
* mental status disorder,
* dementia,
* cognitive impairment,
* intubation,
* tracheostomy,
* need for oxygen therapy due to pre-existing disease,
* patients on home oxygen or ventilator,
* pregnancy,
* recent history of epistaxis or allergy to propofol patients will be excluded.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: GRUP N:(nasal grup: n=60) retrospektif =Patient data will be recorded from the retrospective patient file and archive.
  GRUP H:( high flow grup: n=60)= The patient group with prospective HFNO will be included in the study and their data will be recorded.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-06-14 (Estimated); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-07-25 (Estimated)

PRIMARY OUTCOMES:
Endotracheal intubation rate or complication | 6 month
  proportion of endotracheal intubation or complication

SECONDARY OUTCOMES:
Length of hospital stay | 6 MONTH
  Time in hospital in days

OTHER OUTCOMES:
Patient confort score | 6 month
  Visual scale varying from 0 (no disconfort) to 4 (maximal disconfort)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Thiruvenkatarajan V, Dharmalingam A, Arenas G, Wahba M, Steiner R, Kadam VR, Tran A, Currie J, Van Wijk R, Quail A, Ludbrook G. High-flow nasal cannula versus standard oxygen therapy assisting sedation during endoscopic retrograde cholangiopancreatography in high risk cases (OTHER): study protocol of a randomised multicentric trial. Trials. 2020 May 29;21(1):444. doi: 10.1186/s13063-020-04378-z. PMID 32471494
- [Result] Schumann R, Natov NS, Rocuts-Martinez KA, Finkelman MD, Phan TV, Hegde SR, Knapp RM. High-flow nasal oxygen availability for sedation decreases the use of general anesthesia during endoscopic retrograde cholangiopancreatography and endoscopic ultrasound. World J Gastroenterol. 2016 Dec 21;22(47):10398-10405. doi: 10.3748/wjg.v22.i47.10398. PMID 28058020
- [Result] Cha B, Lee MJ, Park JS, Jeong S, Lee DH, Park TG. Clinical efficacy of high-flow nasal oxygen in patients undergoing ERCP under sedation. Sci Rep. 2021 Jan 11;11(1):350. doi: 10.1038/s41598-020-79798-7. PMID 33432035